CLINICAL TRIAL: NCT04156581
Title: Erector Spinae Plane Block Versus Conventional Analgesia in Complex Spine Surgery: A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Conventional Analgesia in Complex Spine Surgery
Acronym: ESPB-Spine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-1282
Record Dates: First submitted 2019-10-25; First posted 2019-11-07 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESPB with Bupivacaine and Dexamethasone (Active Comparator): 23 complex spine surgery patients will be randomized to receive intraoperative ultrasound-guided bilateral ESPB with 0.375% bupivacaine plus 2 mg preservative free dexamethasone, 25-30 mL total per side according to patient weight.
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone
- ESPB with saline placebo (Placebo Comparator): 23 complex spine surgery patients will be randomized to receive intraoperative ultrasound-guided bilateral ESPB with saline placebo, 25-30 mL total per side according to patient weight.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine is administered typically to reduce sensation in an area. It acts as a nerve block for surgical procedures.
  Other Names: Marcaine
  Arms: ESPB with Bupivacaine and Dexamethasone
Drug: Dexamethasone — Dexamethasone is a corticosteroid that reduces inflammation.
  Other Names: Decadron
  Arms: ESPB with Bupivacaine and Dexamethasone
Other: Saline — Saline is a mixture of NaCl and water that can be used as a placebo.
  Other Names: sodium chloride
  Arms: ESPB with saline placebo

SUMMARY:
Enhanced recovery pathways (ERPs) emphasize evidence-based, multimodal anesthetic and analgesic choices to minimize opioid consumption while providing adequate pain control after surgery. Although ERPs for spine surgery are now being described, few pathways include regional analgesia. The Erector Spinae Plane Block (ESPB) may represent a novel opportunity to incorporate regional analgesia into ERPs for spine surgery. To date, there is minimal data to support the utility of ESPB in spine surgery, and this block has not yet been evaluated in complex spine surgery.

This study seeks to see whether ESPB will reduce opioid consumption and pain scores, and improve patient recovery during the first 24 hours after complex spine surgery when included in a comprehensive ERP.

DETAILED DESCRIPTION:
Lumbar spinal fusion with posterior approach is a moderate-severely painful procedure requiring significant postoperative opioid analgesia (Mathiesen, 2013). There are limited opportunities to use multimodal analgesia (MMA) and regional analgesia after spine surgery. For example, non-steroidal anti-inflammatory drugs are not universally provided, due to concerns regarding bleeding and impaired fusion (Sivaganasan, 2017). Likewise, local anesthetic-based techniques may cause motor weakness and sensory changes which interfere with interpretation of the early postoperative neurological examination.

As in other orthopedic subspecialty surgeries, enhanced recovery pathways (ERPs) are now being described in spine surgery (Wang 2017; Soffin 2018; Soffin 2019a; Ali 2019). Published data emphasizes the importance of opioid-sparing MMA to achieve analgesia and minimize opioid-related side effects. However, with the exception of a report from our group, none include regional analgesia or field blocks as an element of care (Soffin 2019b). Further, comparative research regarding the benefits of regional analgesia within standardized ERPs is lacking for other surgical modalities - even within subspecialties where the evidence base to support such trials is more advanced. These deficits highlight an opportunity to demonstrate the unique advantages of regional analgesia over and above that which can be provided by conventional oral and/or intravenous MMA.

Ultrasound-guided erector spinae plane block (ESPB) may represent a novel opportunity to apply regional analgesia to patients undergoing spine surgery. First described in 2016, ESPB provides analgesia by depositing local anesthetic deep to the erector spinae muscles (Forero 2016). Studies have not completely defined the mechanism of the block, but the target of the local anesthetic has been proposed to be unmyelinated C fibers / sensory cell bodies within the dorsal root ganglia (Ivanusic 2018).

Since its introduction, hundreds of case reports with a wide spectrum of indications have described ESPB as a useful analgesic adjunct for a wide range of indications (Tsui 2019). The feasibility of ESPBs in spine surgery has likewise been suggested in case reports (Almeida 2019; Chin 2019), case series (Melvin 2018; Singh 2018) and retrospective cohort studies (Ueshima 2019). Each conclude significant opioid-sparing capacity and improved NRS pain scores in patients who receive ESPB for a variety of spine surgery procedures.

More recently, results from 2 RCTs describing outcomes after ESPB for lumbar decompression have been reported. In the first, 60 patients were randomized to receive bilateral ESPB or no intervention (Yayik 2019). NRS scores and tramadol consumption were significantly lower in the first 24 hours after surgery, and the time to requesting opioid analgesia was significantly longer in patients were received ESPB. In the second RCT, postoperative morphine consumption was lower in patients who received ESPB compared to patients who did not receive ESPB (Singh, 2019). NRS scores were lower up to 6 hours after surgery in the ESPB group, and patient satisfaction scores were higher.

These preliminary RCTs are promising; however, both suffer from methodological flaws, including lack of power, inadequate blinding, and incomplete standardization of other intra- and post-operative analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Planned primary complex spine surgery: >2 level- lumbar and/or thoraco-lumbar spine fusion with or without decompression
* Planned stand-alone posterior surgical approach
* Able to follow study protocol
* Able to communicate in English (outcome questionnaires validated in English)

Exclusion Criteria:

* Age <18 or >80
* Revision surgery
* BMI > 35
* planned prolonged intubation/intubation overnight on night of surgery
* Unable to communicate in English
* History of chronic pain condition requiring gabapentin/pregabalin/antidepressant medication longer than 3 months
* Opioid tolerance (>60 OME daily for >2 weeks)
* Allergy, intolerance or contraindication to any protocol component/study medication/technique
* Patient refusal of regional analgesia (ESPB)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Soffin, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Certain individual participant data will be available. Individual participant data that underlie the results reported in a future article, after deidentification (text, tables, figures, appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment conducted at the Hospital for Special Surgery between 11/2019 and 6/2022.
Period: Overall Study
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — The age of the participant at the time of enrollment. Measured in years.
  years | 59.13 (18.02) | 57.26 (16.48) | 58.2 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants] — The participant's sex as reported by the patient.
  Participants
    Female | 12 | 16 | 28
    Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The self-reported race of the participant.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 22 | 20 | 42
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — The participants' body mass index at the time of study enrollment.
  kg/m^2 | 25.36 (4.35) | 24.49 (3.55) | 24.93 (3.95)
Weight [Mean (Standard Deviation); unit: kg] — The participants' weight at the time of study enrollment.
  kg | 70.46 (16.31) | 66.23 (12.88) | 68.35 (14.69)
Height [Mean (Standard Deviation); unit: meters] — The participants' height at the time of study enrollment.
  meters | 1.66 (.014) | 1.64 (0.1) | 1.65 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative and Postoperative Opioid Consumption
Description: The total amount of opioid taken during surgery and 24 hours after surgery, measured in morphine milligram equivalent (MME).
Time Frame: 0-24 hours after surgery (intraoperative + immediately after surgery)
Measure: Mean (Standard Deviation); unit: MME/day
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 23 | 23
MME/day | 191 (195.2) | 139.4 (70.5)

2. Secondary Outcome: Numeric Rating Scale Pain at Rest
Description: Measured by Numeric Rating Scale (NRS) pain at rest (The minimum value 0 being 'no pain' and the maximum value 10 being 'as bad as you can imagine').
  Higher scores means a worse outcome.
Time Frame: at baseline (holding area), post anesthesia care unit (PACU) (hour 0), hour 6, 12, and 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 23 | 23
score on a scale
  Pain Scores at Rest at baseline | 2.74 (2.56) | 3.04 (2.2)
  Pain Scores at Rest at PACU (0 hours) | 3.56 (3.93) | 4.15 (4.07)
  Pain Scores at Rest at 6 hours | 3.33 (2.35) | 3.9 (2.49)
  Pain Scores at Rest at 12 hours | 3.19 (2.1) | 3.87 (2.53)
  Pain Scores at Rest at 24 hours | 3.86 (2.1) | 4.05 (1.96)

3. Secondary Outcome: Pain Scores With Physical Therapy
Description: Measured by Numeric Rating Scale (NRS) pain with movement (The minimum value 0 being 'no pain' and the maximum value 10 being 'as bad as you can imagine').
  Higher scores means a worse outcome.
Time Frame: on post-operative physical therapy day 0, 1, and 2
Population: The Number of Participants Analyzed differs from the number of participants assigned to each arm due to lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 21 | 20
score on a scale
  Pain with movement (physical therapy) at POD 0 | 3 (1.41) | 2 (2.45)
  Pain with movement (physical therapy) at POD 1 | 4.29 (2.8) | 3.9 (2.29)
  Pain with movement (physical therapy) at POD 2 | 4.94 (2.95) | 3.53 (2.85)

4. Secondary Outcome: Quality of Recovery
Description: Quality of recovery (QoR) after anesthesia measures the early postoperative health status of patients. QoR15 is the shortened (15 questions) version, each question is scored on the following scales: (Part A: 0 to 10 where 0=none of the time [poor] and 10=all the time [excellent]; Part B: 0 to 10 where 10=none of the time [poor] and 0=all the time [excellent]).
  The total recovery score is scored on the following scale excellent= 136-150, good=122-135, moderate=90-121, and poor=0-89.
  A lower score means a worst outcome.
Time Frame: at baseline (holding area), 24 and 72 hours after surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 22 | 20
score on a scale
  Quality of recovery (QoR) at preop | 101.36 (10.62) | 99.45 (10.53)
  Quality of recovery (QoR) at 24 hours | 69.85 (14.75) | 74.73 (10.22)
  Quality of recovery (QoR) at 72 hours | 79.67 (11.89) | 79.82 (12.53)

5. Secondary Outcome: Opioid Related Side Effects
Description: The Opioid-Related Symptom Distress Scale (ORSDS) is a 4-point scale (minimum = 0 to maximum = 4) that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness). Measured by 10 symptoms on the following scale: did not have symptom = 0, slight = 1, moderate = 2, severe = 3, very severe = 4.
  The total score for each participant was calculated and then the average score for the group was reported.
Time Frame: at 24 hours after surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 18 | 14
score on a scale | 2.56 (0.67) | 2.24 (0.65)

6. Secondary Outcome: Blinding Assessment
Description: Measured by bang blinding index (choose between two treatment arms and provide explanation as to why arm was chosen). The blinding index proposed is scaled to an interval of -1 to 1, 1 being complete lack of blinding, 0 being consistent with perfect blinding and -1 indicating opposite guessing which may be related to unblinding.
  The blinding assessment was completed by the participant, research assistant and anesthesiologist (principle investigator).
Time Frame: at 72 hours after surgery
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 22 | 22
score on a scale
  Bang Blinding Index (participants' response) | .045 [-0.24 to 0.33] | -0.048 [-0.33 to 0.23]
  Bang Blinding Index (research assistant's response) | 0.318 [0.01 to 0.62] | -0.045 [-0.37 to 0.28]
  Bang Blinding Index (anesthesiologist's response) | 0.381 [0.08 to 0.64] | -0.429 [-0.73 to -0.12]

7. Secondary Outcome: Time to First Opioid Use Via Intravenous Administration
Description: Time to pressing opioid use via intravenous administration (IV PCA)
Time Frame: up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 22 | 22
minutes | 237.73 (185.91) | 286.23 (458.77)

8. Secondary Outcome: Time to Opioid Consumption Via Oral Administration
Description: Time to pressing opioid use via oral administration (Oral PCA)
Time Frame: up to 24 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 21 | 23
minutes | 254.62 (360.87) | 141.09 (271.87)

9. Secondary Outcome: Total Opioid Consumption
Description: Measured in morphine milligram equivalent (MME).
Time Frame: 0-12 hours after surgery (intraoperative + immediately after surgery)
Measure: Mean (Standard Deviation); unit: MME/day
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 23 | 23
MME/day | 21.83 (15.42) | 25.48 (18.37)

10. Secondary Outcome: 24 Hours Post-operative Opioid Consumption
Description: The total opioid consumption at 24 hours post-operatively, measured in morphine milligrams equivalent (MME).
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: MME/day
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
Number analyzed (Participants) | 23 | 23
MME/day | 42.9 (31.1) | 47.6 (33.2)

ADVERSE EVENTS:
Time Frame: Adverse events data will be collected over the course of study enrollment and research activities. For this study, adverse events for each participant were assessed from the day of enrollment to the last day of study follow up, post-operative day 3.
Arm/Group | ESPB With Bupivacaine and Dexamethasone | ESPB With Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESPB With Bupivacaine and Dexamethasone (N=23) | ESPB With Saline Placebo (N=23)
Post-operative tachycardia and hypoxia (General disorders) | 0 (0) | 1 (1) — The participant had new-onset tachycardia and hypoxia after surgery, and a CT scan showed that they had segmental and subsegmental pulmonary emboli on both sides in various lobes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04156581/Prot_SAP_000.pdf